CLINICAL TRIAL: NCT01183000
Title: Effects of Closure Versus Non-closure of the Visceral and Parietal Peritoneum at Cesarean Section on Adhesions: A Prospective Randomized Study
Brief Title: Closure of Peritoneum at Cesarean Section and Postoperative Adhesion
Acronym: cs adhesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, ofer gemer, Prof. Ofer Gemer, Barzilai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1789
Record Dates: First submitted 2010-08-08; First posted 2010-08-17 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cesarean Section; Adhesions
Keywords: Formation of adhesions assessed at subsequent cs
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peritoneal closure (Active Comparator)
  Interventions: Procedure: Closure of the peritoneum at cs
- Non closure of the peritoneum (No Intervention)

INTERVENTIONS:
Procedure: Closure of the peritoneum at cs — Injection of 5 mg Marcaine (anesthetic solution) to the leg
  Arms: peritoneal closure

SUMMARY:
Objective: To determine the effect of non-closure of the visceral and parietal peritoneum during Cesarean section on the formation of adhesions.

Study design: A prospective randomized trial of 533 women undergoing primary Cesarean section; 256 were randomized to non closure and 277 to closure of the peritoneum. At a subsequent cesarean,he presence of adhesions and their severity was evaluated at several sites: between the layers of the abdominal wall, between the bladder and the abdominal wall, between bladder and uterus, between the uterus and the abdominal wall, and between the bowels and the pelvic organs. A cumulative adhesion score was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing primary CS

Exclusion Criteria:

* Lack of consent by the patient or an urgent cesarean not allowing time to elicit an informed consent
* Previous pelvic or abdominal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2010-01-16 (Actual); Primary Completion 2010-08-16 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Adhesion score | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gemer, MD, Principal Investigator — Barzili Medical Center
Locations (2):
- Israel (2):
  - Barzilai Medical Center, Ashkelon
  - Barzilay University Medical Center, Ashkelon